CLINICAL TRIAL: NCT04882254
Title: Normothermic Machine Perfusion as Additional Value to Hypothermic Machine Perfusion for Kidney Transplant Outcomes. A Single-centre, Open-label, Randomised, Controlled Trial.
Brief Title: Normothermic Machine Perfusion: an Additional Value for Kidney Transplant Outcomes?
Acronym: APOLLO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Robert Minnee, Transplant surgeon, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APOLLO
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Kidney Transplant Failure; Chronic Kidney Failure
Keywords: Normothermic kidney machine perfusion
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: 1:1 randomised to either intervention arm (normothermic machine perfusion, NMP) or standard-of-care (hypothermic machine perfusion, HMP)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normothermic machine perfusion (Experimental): Additional 2 hours of normothermic machine perfusion of donor kidney with a red cell based perfusate.
  Interventions: Procedure: Normothermic machine perfusion
- Standard-of-care (No Intervention): Standard-of-care, which is hypothermic kidney machine perfusion in the Netherlands.

INTERVENTIONS:
Procedure: Normothermic machine perfusion — Additional 2h of normothermic machine perfusion of the donor kidney with a red cell based perfusate.
  Arms: Normothermic machine perfusion

SUMMARY:
This study is a randomised, controlled, phase II trial to assess the efficacy of 2 hours normothermic machine perfusion (NMP) of extended criteria(EC)-DBD (donation after brain death) and DCD (donation after circulatory death) donor kidneys compared to standard care, which is hypothermic machine perfusion (HMP) only in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* kidney-only transplant
* renal replacement therapy at time of transplant
* receiving standard immunosuppression regimen post-transplant.
* Donation after circulatory death (DCD) Maastricht type III, IV, or V or extended criteria donation after brain death (DBD) donor kidneys.

Exclusion Criteria:

* pre-emptive at time of transplant
* receive a multi-organ or dual kidney transplant
* age donor or recipient below 18 years
* Maastricht type I and II DCD
* donor kidneys preserved on static cold storage (SCS)
* kidneys retrieved after normothermic regional perfusion (NRP)
* Recipient virtual panel reactive antibodies ≥85%
* Recipient for who it is agreed in advance that dialysis after transplant is required, such as in the context of hyperoxaluria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with immediate graft function | 3 months
  Immediate graft function, which is defined as no delayed graft function and/or no primary non-function of the kidney graft.

SECONDARY OUTCOMES:
Duration of delayed graft function | 3 months
estimated glomerular filtration rate (eGFR) trajectory in the first year post-transplant | 1 year
Number of patients with biopsy-proven acute rejection (BPAR) within the first year post-transplant | 1 year
all-cause and death-censored graft survival up to 5 years | 5 years
patient survival up to 5 years | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC Transplant Institute, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin H, Bousnina K, Slagter JS, Fang Y, Cristoferi I, Garrelds IM, Danser AHJ, Reinders MEJ, Minnee RC, Hoogduijn MJ. (Pro)renin, Erythropoietin, Vitamin D and Urodilatin Release From Human Donor Kidneys During Normothermic Machine Perfusion: Predictors of Early Post-Transplant Outcome? Clin Transplant. 2025 May;39(5):e70163. doi: 10.1111/ctr.70163. PMID 40278798
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743
- [Derived] Rijkse E, Bouari S, Kimenai HJAN, de Jonge J, de Bruin RWF, Slagter JS, van den Hoogen MWF, IJzermans JNM, Hoogduijn MJ, Minnee RC. Additional Normothermic Machine Perfusion Versus Hypothermic Machine Perfusion in Suboptimal Donor Kidney Transplantation: Protocol of a Randomized, Controlled, Open-Label Trial. Int J Surg Protoc. 2021 Oct 6;25(1):227-237. doi: 10.29337/ijsp.165. eCollection 2021. PMID 34708171